CLINICAL TRIAL: NCT04571996
Title: Blood-Brain Barrier Penetration of Therapeutic Agents in Human - an Exploratory Repeated Dose Pharmacokinetic Study in Patients With Idiopathic Normal Pressure Hydrocephalus Treated With Cerebroventricular Shunting
Brief Title: Blood-Brain Barrier Penetration of Therapeutic Agents in Human
Acronym: BRIAN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3112012
Record Dates: First submitted 2020-09-25; First posted 2020-10-01 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: CNS Disease
Keywords: Method; Blood Brain Barrier; Penetration; Therapeutics
MeSH Terms: conditions — Central Nervous System Diseases | interventions — Acetaminophen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ODM-104 and Panadol Zapp (Experimental)
  Interventions: Drug: ODM-104; Drug: Paracetamol

INTERVENTIONS:
Drug: ODM-104 — Capsule
Drug: Paracetamol — Rapidly dissolving tablet
  Other Names: Panadol Zapp

SUMMARY:
This is a phase 1, open-label, non-randomized, exploratory, repeated dose PK study performed at a single centre. Up to 6 evaluable subjects are planned. The subjects will receive p.o. doses of ODM-104 for 5-7 days. Single dose of paracetamol will be administered p.o. together with ODM-104 for purposes of comparison.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent (IC) obtained before any study assessments are performed.
2. Sufficient command of the Finnish language to be able to understand the subject information and to communicate with the study personnel.
3. Males and females over 18 years of age.
4. Body mass index (BMI) between 18-30 kg/m2.
5. Idiopathic normal pressure hydrocephalus.
6. Shunt surgery with cerebroventricular catheter placed at least 3 months earlier.
7. Good general health, based on medical history, physical examination and laboratory assessments.
8. Adequate mental status to give informed consent as assessed by the investigator and using the Consortium to Establish a Registry for Alzheimer's Disease (CERAD) neuropsychological battery.
9. Female participants of child-bearing potential and male participants with female partners of child-bearing potential must adhere to a highly effective form of contraception (listed in Section 4.6) from the first study treatment administration until 1 month after the EoS visit.

Exclusion Criteria:

1. Predicted poor compliance with study procedures, restrictions and requirements.
2. Vulnerable subjects (i.e. persons under any administrative or legal supervision).
3. Veins unsuitable for repeated venipuncture or cannulation
4. Evidence of other current clinically significant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolicendocrine, neurological, urogenital or psychiatric disease than iNPH, as judged by the investigator.
5. Type 1 diabetes mellitus.
6. Diagnosis of cancer for which the subject is currently being treated, or for which there is evidence of active disease. Subjects with local prostate cancer or local dermatological tumours, such as basal or squamous cell carcinoma, may be included.
7. Susceptibility to severe allergic reactions, e.g. history of anaphylactic shock due to any reason.
8. Use of medications impacting the metabolism of dopamine, such as other COMT inhibitors (e.g. entacapone), levodopa and monoamine oxidase (MAO) inhibitors (e.g. rasagiline, selegiline), within 4 weeks before the first study drug administration.
9. Any clinically significant abnormalities in screening laboratory test results, vital signs or physical examination findings that might influence the results of the study or cause a health risk for the subject if he/she takes part in the study.
10. Any clinically significant 12-lead ECG abnormality, such as QTcF > 450 ms, after 10 min rest in supine position at the screening visit.
11. Heart rate (HR) < 50 bpm or > 90 bpm, systolic blood pressure (BP) < 90 mmHg or > 160 mmHg, or diastolic BP < 50 mmHg or > 100 mmHg in supine or seated position after 10 min rest at the screening visit.
12. Positive serology to human immunodeficiency virus antibodies (HIVAgAb), hepatitis C virus antibodies (HCVAb) or hepatitis B surface antigen (HBsAg).
13. History of alcohol or drug abuse within the last 5 years, or current regular use of illicit drugs or excessive use of alcohol (regular alcohol drinking of more than 24 units/week for males or 14 units/week for females), or positive breath test for alcohol or positive urine test for drugs of abuse at screening or prior to the first IMP administration.
14. Inability to refrain from consuming caffeine-containing beverages during the stay in the unit.
15. Current use of nicotine-containing products, more than 5 cigarettes or equivalent/day, or inability to refrain from using nicotine-containing products during the stay at the study centre.
16. Pregnant or lactating females.
17. Participation in any other clinical drug study within 2 months before the first IMP administration of this study.
18. Blood donation or loss of significant amount of blood within 2 months prior to the screening visit.
19. Employee or first-degree relative of an employee of the contract research organization (CRST) or Orion.
20. Any other condition that in the opinion of the investigator might interfere with the evaluation of the study results or constitute a health risk for the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Cmax | Daily PK samples during the first and last day of administration from day 1 to day 5-7
  In plasma / CSF
Tmax | Daily PK samples during the first and last day of administration from day 1 to day 5-7
  In plasma / CSF
AUC | Daily PK samples during the first and last day of administration from day 1 to day 5-7
  In plasma / CSF
Cav | Daily PK samples during the first and last day of administration from day 1 to day 5-7
  In plasma / CSF
M/P ratio | Daily PK samples during the first and last day of administration from day 1 to day 5-7
  In plasma / CSF

CONTACTS AND LOCATIONS:
Overall Officials: Orion Pharma Clinical study director, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- CRST Turku, Turku, Finland